CLINICAL TRIAL: NCT03980314
Title: A Randomized, Double-Blind, Parallel, Phase 1 Study to Compare the Pharmacokinetics of BMSCHO1-Nivolumab Process D to Nivolumab Process C After Complete Resection of Stage IIIa/b/c/d or Stage IV Melanoma
Brief Title: A Study to Compare Nivolumab Drug Product Process D to Nivolumab Drug Product Process C in Participants With Stage IIIa/b/c/d or Stage IV Melanoma After Complete Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-8FC; 2018-002993-38 (EudraCT Number)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Process C) (Active Comparator)
  Interventions: Drug: Nivolumab
- Arm B (Process D) (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to compare the drug levels, immunogenicity and safety of Nivolumab Process D to Nivolumab Process C after complete resection of stage IIIa/b/c/d or stage IV melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIa/b/c/d or stage IV melanoma
* Complete resection of Stage III disease that is documented on the surgical and pathology reports or complete resection of Stage IV disease with margins negative for disease that is documented on the pathology report
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Prior malignancy active within the previous 3 years, except for locally curable cancers that have been apparently cured
* Any significant acute or chronic medical illness that is uncontrolled
* History of ocular/uveal melanoma
* Active, known or suspected autoimmune disease
* Systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent, are permitted in the absence of active autoimmune disease.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve in one dosing interval (AUC[TAU]) (336 h) | Over the dosing interval at Week 1 and Week 17

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Over the dosing interval at Week 1 and Week 17
Observed serum concentration at the end of a dosing interval (Ctau) | Over the dosing interval at Week 1 and Week 17
Time of maximum observed plasma concentration (Tmax) | Over the dosing interval at Week 1 and Week 17
Number of Participants With Positive Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) | Through Week 51 Day 1
Number of Participants With Serious Adverse Events (SAEs) | Up to 65 weeks
Number of Participants With Adverse Events leading to Discontinuation | Up to 65 weeks
Number of Participants With Adverse Events (AEs) | Up to 65 weeks
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 65 weeks
Number of Participants with AEs leading to death | Up to 65 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (37):
- United States (4):
  - Local Institution - 0006, Hartford, Connecticut
  - Local Institution - 0008, Minneapolis, Minnesota
  - Local Institution - 0035, Charlotte, North Carolina
  - Local Institution - 0043, Pittsburgh, Pennsylvania
- Local Institution - 0046, Buenos Aires, Argentina
- Local Institution - 0001, Wollstonecraft, New South Wales, Australia
- Brazil (6):
  - Local Institution - 0036, Ijuí, Rio Grande do Sul
  - Local Institution - 0037, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0039, Barretos, São Paulo
  - Local Institution - 0038, Cerqueira César, São Paulo
  - Local Institution - 0040, São José do Rio Preto, São Paulo
  - Local Institution - 0041, Rio de Janeiro
- Local Institution - 0013, Edmonton, Canada
- Chile (4):
  - Local Institution - 0024, Independencia, Santiago Metropolitan
  - Local Institution - 0045, Santiago, Santiago Metropolitan
  - Local Institution - 0023, Santiago, Santiago Metropolitan
  - Local Institution - 0022, Santiago
- France (3):
  - Local Institution - 0009, Marseille
  - Local Institution - 0010, Nantes
  - Local Institution - 0011, Paris
- Ireland (2):
  - Local Institution - 0018, Wilton, CORK
  - Local Institution - 0032, Dublin
- Italy (3):
  - Local Institution - 0014, Bergamo
  - Local Institution - 0015, Padua
  - Local Institution - 0016, Siena
- Mexico (3):
  - Local Institution - 0034, Tlalpan, Mexico City
  - Local Institution - 0033, Monterrey, Nuevo León
  - Local Institution - 0031, San Pedro Garza García, Nuevo León
- New Zealand (3):
  - Local Institution - 0005, Auckland
  - Local Institution - 0004, Christchurch
  - Local Institution - 0003, Wellington
- Local Institution - 0017, Warsaw, Poland
- Local Institution - 0030, Timișoara, Romania
- Spain (4):
  - Local Institution - 0029, Badalona-barcelona
  - Local Institution - 0026, Madrid
  - Local Institution - 0027, Madrid
  - Local Institution - 0028, Málaga

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm